CLINICAL TRIAL: NCT03212404
Title: A Phase 1, Open-label, Multicenter, Dose-escalation Study of CK-301 Administered Intravenously as a Single Agent to Subjects With Advanced Cancers
Brief Title: Phase 1 Study of CK-301 (Cosibelimab) as a Single Agent in Subjects With Advanced Cancers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Checkpoint Therapeutics, Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CK-301-101
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Small Cell; Malignant Mesothelioma, Advanced; Head and Neck Cancer; Melanoma; Merkel Cell Carcinoma; Renal Cell Carcinoma; Urothelial Carcinoma; Classical Hodgkin Lymphoma; Cutaneous Squamous Cell Carcinoma; Non Hodgkin Lymphoma; Endometrial Cancer
Keywords: Cancer; PD-L1; PDL1; PD-1; PD1; Solid tumors; Anti PD-L1; Non-small cell lung cancer, NSCLC; CK-301; CSCC; Skin cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Small Cell; Mesothelioma, Malignant; Head and Neck Neoplasms; Melanoma; Carcinoma, Merkel Cell; Carcinoma, Renal Cell; Carcinoma, Transitional Cell; Lymphoma, Non-Hodgkin; Endometrial Neoplasms; Neoplasms; Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CK-301 (cosibelimab) (Experimental): Part 1 - Dose Escalation; Part 2 - Dose Expansion
  Interventions: Drug: CK-301 (cosibelimab)

INTERVENTIONS:
Drug: CK-301 (cosibelimab) — CK-301 will be administered in periods of 28-day cycles.

SUMMARY:
CK-301 (cosibelimab) is a fully human monoclonal antibody of IgG1 subtype that directly binds to Programmed Death-Ligand 1 (PD-L1) and blocks its interactions with the Programmed Death-1 (PD-1) and B7.1 receptors. The primary objectives of this study are to assess the safety, tolerability and efficacy of CK-301 when administered intravenously as a single agent to subjects with selected recurrent or metastatic cancers.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1, open-label, multicenter, dose-escalation study of CK-301 (cosibelimab), a fully human monoclonal IgG1 antibody targeting PD-L1. The study will consist of 3 periods: Screening (up to 28 days), Treatment (28-day cycles), and Follow-up (up to 6 months of visits with survival follow-up for select cohorts). Following the dose escalation portion of the study, additional evaluable subjects may be included in order to further characterize safety and efficacy at selected doses and/or in specific patient sub-groups.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Male or female subjects aged greater than or equal to 18 years.
* For NSCLC: Histologically or cytologically confirmed diagnosis of unresectable recurrent or metastatic non-small cell lung cancer.
* For CRC: Histologically confirmed diagnosis of recurrent or metastatic colorectal cancer assessed as microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR).
* For EC: Histologically or cytologically confirmed advanced, recurrent or metastatic endometrial carcinoma.
* For cSCC: Histologically confirmed diagnosis of unresectable or metastatic cutaneous squamous cell carcinoma not amenable to local therapy.
* For SCLC: Histologically or cytologically confirmed diagnosis of unresectable small cell lung cancer.
* For MPM: Histologically or cytologically confirmed diagnosis of unresectable malignant pleural or peritoneal mesothelioma.
* For HNSCC: Histologically or cytologically confirmed diagnosis of recurrent or metastatic HNSCC (oral cavity, pharynx, larynx), stage III/IV and not amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy).
* For MEL: Histologically confirmed diagnosis of unresectable Stage III or metastatic melanoma not amenable to local therapy (excluding uveal or ocular melanoma).
* For MCC: Histologically confirmed diagnosis of metastatic Merkel cell carcinoma not amenable to local therapy.
* For RCC: Histologically confirmed diagnosis of renal cell carcinoma (with clear cell component) with advanced or metastatic disease that is not amenable to cure by surgery or other means.
* For UC: Histologically or cytologically documented locally advanced or metastatic transitional cell carcinoma of the urothelium (including renal pelvis, ureters, urinary bladder, urethra) not amenable to cure by surgery or other means.
* For HL: Histologically confirmed primary diagnosis of classical Hodgkin's lymphoma.
* For B-cell NHL: Histologically confirmed diagnosis of non-Hodgkin lymphoma.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at trial entry and an estimated life expectancy of at least 3 months
* Must have at least one measurable lesion based on RECIST 1.1.
* Have provided a formalin fixed tumor tissue sample from a biopsy of a tumor lesion either at the time of or after the diagnosis of metastatic disease has been made AND from a site not previously irradiated.
* Adequate hematological, hepatic and renal function as defined in the protocol.
* Effective contraception for both male and female subjects if the risk of conception exists.
* Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
* Concurrent treatment with a non-permitted drug.
* History of severe hypersensitivity reactions to other monoclonal antibodies.
* Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast, or localized prostate cancer.
* Chemotherapy, radioactive, biological cancer therapy, or tyrosine kinase inhibitor (TKI) therapy, within four weeks prior to the first dose of study drug, or who has not recovered to NCI CTCAE Grade 1 or better from the AEs due to cancer therapeutics administered more than four weeks earlier.
* Significant acute or chronic infections as defined in the protocol.
* Active or history of interstitial lung disease (ILD), or has had a history of pneumonitis that has required oral or IV steroids.
* Active or suspected autoimmune disease or a documented history of autoimmune disease.
* Known current drug or alcohol abuse.
* Underlying medical conditions that will make the administration of study drug hazardous or obscure the interpretation of toxicity determination or adverse events.
* Use of other investigational therapy within 28 days before study drug administration.
* Pregnant or breastfeeding.
* Uncontrolled or significant cardiovascular disease.
* Psychiatric illness or social situation that would preclude study compliance.
* Receipt of live, attenuated vaccine within 28 days prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | Up to 4 weeks
Number of subjects with Treatment-Emergent Adverse Events according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03 (or most current version) | Screening through 4 weeks after study completion, an average of 6 months
Confirmed Objective Response Rate (ORR) as per Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) | Part 2 Only: Average of 6 months

SECONDARY OUTCOMES:
Confirmed Best Overall Response (BOR) as per Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) | Every 8 weeks for first 32 weeks, then 12 weeks through study completion, an average of 6 months
Duration of Response (DoR) as per Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) | Every 8 weeks for first 32 weeks, then 12 weeks through study completion, an average of 6 months
Objective response rate and duration of response (DOR) based on Modified RECIST 1.1 for immune based therapeutics | Part 2 Only: Every 8 weeks for first 32 weeks, then 12 weeks through study completion, an average of 6 months
Overall Survival (OS) | Part 2 Only: Every 8 weeks for first 32 weeks, then 12 weeks through study completion, an average of 6 months
Pharmacokinetic parameter: AUC (0-t) of CK-301 | Baseline up to 12 weeks after study completion, an average of 6 months
Pharmacokinetic parameter: AUC (0-infinity) of CK-301 | Baseline up to 12 weeks after study completion, an average of 6 months
Pharmacokinetic parameter: Cmax of CK-301 | Baseline up to 12 weeks after study completion, an average of 6 months
Pharmacokinetic parameter: Tmax of CK-301 | Baseline up to 12 weeks after study completion, an average of 6 months
Pharmacokinetic parameter: T(1/2) of CK-301 | Baseline up to 12 weeks after study completion, an average of 6 months
Number of subjects with anti-CK-301 antibodies | Baseline up to 12 weeks after study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Locations (46):
- Australia (8):
  - Research Site, Wollongong, New South Wales
  - Research Site, Benowa, Queensland
  - Research Site, Buderim, Queensland
  - Research Site, Greenslopes, Queensland
  - Research Site, South Brisbane, Queensland
  - Research Site, Woolloongabba, Queensland
  - Research Site, Box Hill, Victoria
  - Research Site, Malvern, Victoria
- France (5):
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Grenoble
  - Research Site, Lyon
  - Research Site, Nice
- Research Site, Christchurch, New Zealand
- Poland (5):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Warsaw
- Russia (8):
  - Research Site, Chelyabinsk
  - Research Site, Kazan'
  - Research Site, Murmansk
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Tyumen
  - Research Site, Volgograd
- South Africa (5):
  - Research Site, Cape Town
  - Research Site, George
  - Research Site, Port Elizabeth
  - Research Site, Pretoria
  - Research Site, Soweto
- Spain (7):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, San Cristóbal de La Laguna
  - Research Site, Seville
  - Research Site, Valencia
- Thailand (4):
  - Research Site, Hat Yai, Changwat Songkhla
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Khon Kaen
- Ukraine (3):
  - Research Site, Chernivtsi
  - Research Site, Kharkiv
  - Research Site, Sumy

REFERENCES:
- [Derived] Clingan P, Ladwa R, Brungs D, Harris DL, McGrath M, Arnold S, Coward J, Fourie S, Kurochkin A, Malan DR, Mant A, Sharma V, Shue H, Tazbirkova A, Berciano-Guerrero MA, Charoentum C, Dalle S, Dechaphunkul A, Dudnichenko O, Koralewski P, Lugowska I, Montaudie H, Munoz-Couselo E, Sriuranpong V, Oliviero J, Desai J. Efficacy and safety of cosibelimab, an anti-PD-L1 antibody, in metastatic cutaneous squamous cell carcinoma. J Immunother Cancer. 2023 Oct;11(10):e007637. doi: 10.1136/jitc-2023-007637. PMID 37848259